CLINICAL TRIAL: NCT04587011
Title: A Phase 1 Clinical Trial to Explore Pharmacokinetics, Pharmacodynamics and Safety After Twice-daily Dosing of Tegoprazan Tablets in Healthy Subjects
Brief Title: A Study to Explore Pharmacokinetics/Pharmacodynamics and Safety of Tegoprazan BID Dosing in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IN_APA_119
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- T1 (Experimental): Tegoprazan A mg or placebo
  Interventions: Drug: Tegoprazan dose A or placebo
- T2 (Experimental): Tegoprazan B mg or placebo
  Interventions: Drug: Tegoprazan dose B or placebo
- T3 (Experimental): Tegoprazan C mg or placebo
  Interventions: Drug: Tegoprazan dose C or placebo
- T4 (Experimental): Tegoprazan D mg or placebo
  Interventions: Drug: Tegoprazan dose D or placebo

INTERVENTIONS:
Drug: Tegoprazan dose A or placebo — Tegoprazan A mg or placebo taken orally twice daily for 3 days.
  Arms: T1
Drug: Tegoprazan dose B or placebo — Tegoprazan B mg or placebo taken orally twice daily for 3 days.
  Arms: T2
Drug: Tegoprazan dose C or placebo — Tegoprazan C mg or placebo taken orally twice daily for 3 days.
  Arms: T3
Drug: Tegoprazan dose D or placebo — Tegoprazan D mg or placebo taken orally twice daily for 3 days.
  Arms: T4

SUMMARY:
The main purpose of this study is to explore the pharmacokinetics, pharmacodynamics and safety after twice-daily dosing of tegoprazan tablets in healthy subjects.

DETAILED DESCRIPTION:
* To explore the pharmacokinetics, pharmacodynamics and safety in accordance with the dose escalation when tegoprazan is given orally twice daily for 3 days in healthy subjects.
* To compare the pharmacodynamics and safety of tegoprazan oral administration and esomeprazole infusion for 24 hours

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 19 to 45(inclusive) years at screening.
* Subjects with body mass index (BMI) in the range of 18.5 kg/m^2 to 28.0 kg/m^2(inclusive)
* Subjects who voluntarily agreed to participate in the study after being fully informed of the purpose, content, and characteristics of the investigational product(IP) prior to the study participation.

Exclusion Criteria:

1. Past medical history

   * Subjects who are determined by the investigator to have clinically significant history or disease related to the liver, kidney, digestive system, respiratory system, musculoskeletal system, endocrine system, neuropsychiatric system, hemato-oncology system, urinary system and cardiovascular system including cardiac arrhythmia.
   * Subjects who are determined by the investigator to have past history of gastrointestinal diseases (ex.: gastritis, GERD, Crohn's disease, ulcers etc.) or abdominal surgery (except simple appendectomy or herniotomy) that may affect the IP absorption.
2. Diagnostic test and electrocardiogram (ECG)

   * If H. pylori test result is positive at screening
   * If the AST or ALT value is more than 1.25 times the upper limit of normal under the screening test
   * If the total bilirubin value is more than 1.5 times the upper limit of normal under the screening test
   * If the eGFR calculated by CKD-EPI formula is less than 80 mL/min at screening
   * Subjects showing clinically significant abnormalities on ECG at screening
3. Allergy and drug abuse

   * Subjects who are hypersensitive to the investigational product or its active ingredient and any other medications (aspirin, antibiotics etc.)
   * Subjects with history of substance abuse or positive results from drug screening test.
4. Contraindicated drugs/foods

   * Subjects who have been taking any medications (including herbal medicines) or on an abnormal diet (ex: consuming more than 1L of grapefruit juice per day, large amounts of garlic, broccoli and kale, etc.) that can affect the absorption, distribution, metabolism and excretion of the IP within 28 days from the first IP administration date
   * Subjects who took any prescription drugs(ETC) or any over-the-counter drugs(OTC) within 10 days from the first IP administration date
   * Subjects who participated in other clinical trials or bioequivalence test and received other investigational product within 6 months from the first day of the IP administration (allowed to participate only if the other investigational product(s) was(were) not taken)
5. Blood donation and transfusion

   * Subjects who donated whole blood within 60 days from the first day of the investigational product administration
   * Subjects who received blood transfusion or made apheresis blood donation within 30 days from the first day of the IP administration
6. Pregnancy, Breastfeeding, and Contraception

   * Women who are pregnant, breast-feeding or have positive result on pregnancy test.
   * Subjects who are unable to use medically proven dual contraceptive methods or medically acceptable contraceptive method (intrauterine device with proven pregnancy failure rate, concurrent use of physical barrier method and spermicide, vasectomy, tubectomy/ligation, and hysterectomy, etc.) by the subject or spouse or partner from the screening date to 30 days after the last IP administration date.
7. Others

   * Subjects whose weekly alcohol intake exceeds 30g/day in the last 4 weeks prior to the screening visit or found positive on alcohol test
   * Subjects who smoke more than 10 cigarettes/day per week over the last 4 weeks prior to the screening visit
   * Subjects with caffeine consumption of more than 400mg/day per week over the last 4 weeks prior to the screening visit
   * Subjects with clinically significant findings that the investigator determined to be unqualified for participation in the clinical trial

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics Evaluation | Up to 24 hours
  Cmax of Tegoprazan and M1
Pharmacokinetics Evaluation | Up to 24 hours
  AUC0-t of Tegoprazan and M1
Pharmacokinetics Evaluation | Up to 24 hours
  AUC0-∞ of Tegoprazan and M1
Pharmacokinetics Evaluation | Up to 24 hours
  Tmax of Tegoprazan and M1
Pharmacokinetics Evaluation | Up to 24 hours
  t1/2β of Tegoprazan and M1
Pharmacokinetics Evaluation | Up to 24 hours
  CL/F of Tegoprazan
Pharmacokinetics Evaluation | Up to 24 hours
  Vd/F of Tegoprazan
Pharmacokinetics Evaluation | Up to 24 hours
  Css,max of Tegoprazan and M1
Pharmacokinetics Evaluation | Up to 24 hours
  Css,min of Tegoprazan and M1
Pharmacokinetic Evaluation | Up to 24 hours
  Css,avg of Tegoprazan and M1
Pharmacokinetics Evaluation | Up to 24 hours
  AUC48-72h of Tegoprazan and M1
Pharmacokinetics Evaluation | Up to 24 hours
  Tmax,ss of Tegoprazan and M1
Pharmacokinetics Evaluation | Up to 24 hours
  t1/2β,ss of Tegoprazan and M1
Pharmacokinetics Evaluation | Up to 24 hours
  CLss/F of Tegoprazan
Pharmacokinetics Evaluation | Up to 24 hours
  Vdss/F of Tegoprazan

SECONDARY OUTCOMES:
Pharmacodynamics Evaluation | 24 hours
  Mean pH
Pharmacodynamics Evaluation | 24 hours
  Median pH
Pharmacodynamics Evaluation | 24 hours
  TpH>4(%)
Pharmacodynamics Evaluation | 24 hours
  TpH>6(%)
Pharmacodynamics Evaluation | 24 hours
  Basal pH
Pharmacodynamics Evaluation | 24 hours
  Δ TpH>4(%)
Pharmacodynamics Evaluation | 24 hours
  Δ TpH>6(%)
Pharmacodynamics Evaluation | 24 hours
  Δ mean pH
Pharmacodynamics Evaluation | 24 hours
  Δ median pH

CONTACTS AND LOCATIONS:
Overall Officials: Jong Lyul Kim, MD, PhD, Principal Investigator — Inje University
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea